CLINICAL TRIAL: NCT04119245
Title: Evaluation of the Efficiency of I-gel Supraglottic Airway Device in Mechanical Ventilation in Supine and Lateral Decubitus Position in Obese Patient;Prospective Observational Study
Brief Title: Efficiency of I-gel Supraglottic Airway Device in Supine and Lateral Decubitus Position in Obese Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-12-2019
Record Dates: First submitted 2019-08-03; First posted 2019-10-08 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Obesity, Airway
Keywords: obesity; Igel; suraglotic device
MeSH Terms: conditions — Obesity; Ige Responsiveness, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): after induction of general anesthesia, a proper size of Igel will be inserted after compelete muscle relaxation. In order to confirm proper positioning of the I-gel,a fiberoptic bronchoscope will be pass through the device and pushed forward up to1 cm proximal to it to obtain a glottic view, leak airway pressure test will be done.
  Afterwards the same patient will be placed in the lateral decubitus position ,confirmation of I-gel position using fiberoptic bronchoscope will be done and recorded.The leak air way pressure test will be done as previously done in supine position and recorded.
  The patient will be returned to supine position.
  Interventions: Device: I-gel supraglottic airway device

INTERVENTIONS:
Device: I-gel supraglottic airway device — After induction of general anesthesia, we will measure the Oropharyngeal leak airway pressure during controlled ventilation in supine and in positions after insertion of I-gel.

SUMMARY:
Obesity is linked to many complications of respiratory care which are directly related to the obstructive apnea syndrome: difficult airway management including difficult mask ventilation, difficult intubation and obstruction of the upper airway.

I gel which is a non inflatablesupraglottic airway device with a gastric channel is gaining popularity in anesthesia practice because of its ease of insertion and stable positioning.

There are many studies evaluating I-gel for airway managment during different head and necks position ,in prone and lateral position showing both successeful results. Morover, it was evaluated during spontanous and mechanically ventilated patients.

There are limited number of studies evaluating the efficacy of I- gel in mild to moderate obese patients.

The primary aim of this study is to Measure the oropharyngeal airway leak pressure in both supine and lateral position and to determine laryngeal glottic view grade by the fibreoptic bronchoscope.

DETAILED DESCRIPTION:
prospective observational cohort study. Induction of anethesisa will be started after pre-oxygenating the patient for 3min , with administerating Propofol (2mg/kg)(lean body weight)), Fentanyl (2μg/kg) and Atracurium (0.5mg/kg)(based on ideal body weight.The patient will to be ventilated by a 100% oxygen and 1.2% isoflurane with fresh gas flow 6L/min for 5 min.immediately after induction heart rate , blood pressure and oxygen saturation will be recorded.

A proper sized I-gel according to the patient's weight and manifacturer instructions (Intersurgical Ltd, UK) ( 4 or 5 adult sizeI-gel) will be lubricated with a water based lubricant from the front and back sides of the device, will be inserted after compelete muscle relaxation (Train of four = zero) In case of insertion problem various adjuvant manoeuvres will be used such as such as head flexion or extension, or slightly pulling or pushing the device. Any additional manoeuvres will be recorded. If insertion or ventilation fails three times in succession, Endotracheal tube will be immediately inserted and the patient will be excluded from the study. The number of excluded cases will be recorded The circut will be connected to the device,Capnograph will be attached and end tidal carbon dioxide will be recorded.

The ventilator parameters will be set with tidal volume (4-6 ml/kg) at a respiratory rate(12-15 breath/min) to maintain ETCO2 from 30-35 mmHg.

Anaethesia will be maintanied by a mixture of 50% oxygen and 50% medical air,Isoflurane 1.2% and Atracurium (0.01 mg/kg) will be given according to train of four . Analgesia of pethidine 100mg IV will be given as intraoperative analgesia.

In order to confirm proper positioning of the I-gel,a fiberoptic bronchoscope will be pass through the device and pushed forward up to1 cm proximal to it to obtain a glottic view.

Afterwards the same patient will be placed in the lateral decubitus position.Blood pressure,Heart rate ,Oxygen saturation and End tidal CO2 will be recorded immedialy. After confirming proper ventilation as before ,confirmation of I-gel position using fiberoptic bronchoscope will be done and recorded.The leak air way pressure test will be done as previously done in supine position and recorded.

The patient will be returned to supine position where a proper size Orogastric tube will be inserted.The surgery can be started and Heamodynamics and ventilation will be monitored.

By the end of the surgery the patient will be reversed from general anaesthesia by administrating Neostigmine (0.04mg/kg) and Atropine (0.01mg/kg). intravenously at (TOF=3) and the I-gel will be removed at the end.The presence of blood on the I-gel device, or the occurrence of any complications, will be recorded.

The patient will be transfered to the post operative care unit

ELIGIBILITY:
Inclusion Criteria:

BMI: ≥30 - <40. Surgery: short time procedures >60 minutes and ≤. 120 minutes

Exclusion Criteria:

Patientswith neck or upper airway pathologies or other contraindications to supraglottic decives.

Patients at risk of stomach contents regurge e.g. pregnant ,GIT Ulcer, Symptomatic reflux disease or Hiatus hernia ...etc Patients with risk of pulmonary aspiration e.g. Full stomach or incompetent gastro-oesophageal sphincter.

History of gastric band or gastric bypass surgeries. Pregnant females. Laparotomy or laparoscopic procedures. Obstructive sleep apnea Patients with risk of bleeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
comparison between supine and lateral Oropharyngeal leak airway pressure | 1 minute
  Oropharyngeal leak airway pressure during controlled ventilation in supine position after insertion of I-gel by one minute and n lateral position after one minute from setting patient in lateral postion.

SECONDARY OUTCOMES:
Swallowing | 5 hours
  The presence of swallowing difficulties, are questioned preoperatively and 5H postoperatively.
Hoarseness | 5 hours
  The presence of Hoarseness is questioned preoperatively and 5H postoperatively.
Nausea and vomiting | 5 hours
  The presence of nausea and vomiting are questioned preoperatively and 5H postoperatively.
fiberoptic view in supine position | 1 minute
  4 points: only vocal cords can be seen, 3 points: vocal cords and posterior epiglottis can be seen, 2 points: vocal cords and anterior epiglottis can be seen, 1 Point: Vocal cords cannot be seen.
fiberoptic view in lateral position | 1 minute
  4 points: only vocal cords can be seen, 3 points: vocal cords and posterior epiglottis can be seen, 2 points: vocal cords and anterior epiglottis can be seen, 1 Point: Vocal cords cannot be seen.
number of failed attempts of insertion | 1 minutes
  I-gel insertion was facilitated by head flexion or extension, or slightly pulling or pushing the device in case of insertion problem. If insertion or ventilation fails three times in succession, Endotracheal tube would immediately inserted and the patient was excluded from the study. The number of excluded cases were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, M.D., Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bamgbade OA, Macnab WR, Khalaf WM. Evaluation of the i-gel airway in 300 patients. Eur J Anaesthesiol. 2008 Oct;25(10):865-6. doi: 10.1017/S0265021508004511. Epub 2008 Jun 6. No abstract available. PMID 18534042
- [Background] Sanuki T, Uda R, Sugioka S, Daigo E, Son H, Akatsuka M, Kotani J. The influence of head and neck position on ventilation with the i-gel airway in paralysed, anaesthetised patients. Eur J Anaesthesiol. 2011 Aug;28(8):597-9. doi: 10.1097/EJA.0b013e32834698f4. PMID 21505345
- [Background] Saracoglu KT, Demir A, Pehlivan G, Saracoglu A, Eti Z. Analysing the efficacy of the I-gel supraglottic airway device in the supine and lateral decubitus positions. Anaesthesiol Intensive Ther. 2018;50(4):259-262. doi: 10.5603/AIT.a2018.0028. Epub 2018 Sep 17. PMID 30221337